CLINICAL TRIAL: NCT06062797
Title: Improving Patient Understanding in the Preoperative Informed Consent Process of Trauma Patients Using a Mixed Reality Viewer
Brief Title: Improving Patient Understanding in Preoperative Informed Consent Process of Trauma Patients Using a Mixed Reality Viewer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Konstantin Wehrkamp, Principal Investigator, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0936
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Distal Radius Fractures; Ankle Fractures; Proximal Humeral Fracture
Keywords: Distal Radius Fracture; Proximal Humeral Fracture; Ankle Fracture; Mixed Reality; Patient Education; Informed Consent; Patient Satisfaction
MeSH Terms: conditions — Wrist Fractures; Ankle Fractures; Shoulder Fractures; Patient Satisfaction | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mixed Reality (Experimental): Fracture visualization via Mixed Reality Viewer
  Interventions: Device: Mixed Reality Viewer
- X-ray or CT scan (Active Comparator): Fracture visualization via X-ray or CT scan
  Interventions: Device: X-ray or CT scan

INTERVENTIONS:
Device: Mixed Reality Viewer — The Mixed Reality Viewer from Brainlab (Germany) enables the visualization of the fracture via a 3D hologram. In contrast to virtual reality, where the user is in a completely virtual world, the user of the mixed reality viewer sees the 3D hologram implemented in his real environment.
  Arms: Mixed Reality
Device: X-ray or CT scan — X-ray or CT scan enables the visualization of the fracture in 2D.
  Arms: X-ray or CT scan

SUMMARY:
This clinical trial aims to compare a Mixed Reality Viewer in the preoperative informed consent process to standard fracture visualization. The participants population are patients with an indication for surgery of a distal radius fracture, upper ankle fracture or proximal humerus fracture using plate osteosynthesis.

The main questions aim to answer are:

* Does the use of the Mixed Reality Viewer improve patient understanding?
* Does the use of the Mixed Reality Viewer improve patient satisfaction?
* Does the use of the Mixed Reality Viewer reduce patient preoperative anxiety?

Participants will have their fracture presented via the Mixed Reality Viewer. Researchers will compare standard fracture imaging using X-ray or CT scans to see if there is any difference in understanding, satisfaction and anxiety.

DETAILED DESCRIPTION:
In everyday clinical practice, patients receive a verbal explanation of their medical condition, optional treatment options, and information about the benefits, risks and complications of surgery during preoperative education. To visualize the respective fractures to the patients, they are shown using X-rays, CT scans or MRI images. However, these images are often difficult to understand without prior medical knowledge.

A better understanding of the fracture by the patients and a more comprehensible visualization of the operations can lead to better informed consent between the patients and the doctor. Consequential benefits for treatment and postoperative follow-up may follow.

The investigators hypothesis is that fracture visualization using a Mixed Reality Viewer can generate higher fracture understanding in patients. As a result of better education, this visualization method could lead to higher patient satisfaction and anxiety reduction.

Patients with an indication for surgery of a distal radius fracture, upper ankle fracture or proximal humerus fracture using plate osteosynthesis are randomized into the intervention group or the control group. Both study groups watch verbal education via a recorded video. The intervention group afterward receives a fracture visualization via mixed reality glasses. The control group receives fracture visualization via X-ray or CT scan.

In both the intervention group and the control group, the type of fracture, the extent of the fracture, the surgical method, and the benefits and risks of the surgery are explained to the patients during the visualization.

After the explanation is completed, patients are asked to complete a questionnaire regarding satisfaction and fracture understanding.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgery of a distal radius fracture, upper ankle fracture, or proximal humerus fracture using plate osteosynthesis
* Age ≥ 18 years old
* Existing signed confirmation of participation in the study
* Ability to understand a German interview and questionnaire

Exclusion Criteria:

* Epilepsy
* Patients with mental limitations (e.g. dementia) or severe visual impairments that prevent informed consent emergency surgery
* Age < 18 or > 80 years old
* Inability to understand a German interview and questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Understanding | Measurement is assessed via a questionnaire immediately after the procedure.
  A questionnaire is used to determine the patients' level of understanding via content-related questions about their specific fractures. Patients answer questions on a 6-point Likert scale, with higher scores indicating better outcome.
Patient Satisfaction with the educational process assessed by the 6-point Likert scale | Measurement is assessed via a questionnaire immediately after the procedure.
  A questionnaire is used to determine the patient's satisfaction with the educational process. Patients answer questions on a 6-point Likert scale, with higher scores indicating better outcome.
Patient Preoperative Anxiety | Measurement is assessed via a questionnaire immediately after the procedure.
  A questionnaire is used to determine the patient's anxiety regarding their upcoming surgical procedure. Patients answer the question on a 10-point Likert scale, with higher scores indicating worse outcome..

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Gilbert, PD Dr. med, Study Director — LMU Munich
Locations (1):
- Department of Orthopaedics and Trauma Surgery, Musculoskeletal University Center Munich (MUM), University Hospital, LMU Munich, Munich, Bavaria, Germany